CLINICAL TRIAL: NCT05935982
Title: Preliminary Implementation and Development of an Enjoyable Virtual Reality Exercise Program for the Prevention of Cardiometabolic Disease Among Children With Disabilities in School Settings
Brief Title: Virtual Reality Exercise in a Community Highschool for Children With Disabilities
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Byron Lai, Assistant Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-300011314; P50MD017338 (NIH)
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Results first posted 2025-03-14 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Disability Physical; Developmental Disability; Physical Inactivity
MeSH Terms: conditions — Developmental Disabilities; Sedentary Behavior | interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality exercise program in special physical education (Experimental): During normal special physical education hours, participants will be provided with a virtual reality headset and exercise games and be prescribed to exercise at a moderate intensity.
  Interventions: Behavioral: Virtual reality exercise
- Virtual reality exercise program at home (Active Comparator): Participants will be provided with a virtual reality headset and exercise games and be prescribed to exercise at a moderate intensity at home.
  Interventions: Behavioral: Virtual reality exercise

INTERVENTIONS:
Behavioral: Virtual reality exercise — During school special physical education, participants will be asked to exercise using a virtual reality exercise headset, that will be adapted for arm use. Participants will asked to be seated during gameplay. Heart rate will be monitored and recorded during exercise.

SUMMARY:
The purpose of this study is to work with a community engagement group to develop and pilot a protocol for a virtual reality exergaming program for children with special needs at a high school.

DETAILED DESCRIPTION:
A virtual reality exercise program will be run during school special physical education hours at a public high school. The program will be implemented by a person with cerebral palsy. The exercise will include rhythmic movement to music and fitness games.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in school special physical education or self-reported disability
* Note from physician permitting participation in moderate intensity exercise or cleared for sport participation through physical examination that was on file by the school
* Ability to communicate in English (or a caregiver)

Exclusion Criteria:

* Complete blindness or deafness
* Condition that may make participation unsafe

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Byron Lai, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Children's Hospital of Alabama, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants self-selected their exercise setting. One participant signed a digital consent form and chose the school setting, but voluntary withdrew prior to the baseline data collection.
Groups:
- School Based: Participants were asked to exercise on site for 25 minutes 3 times a week during study hall for 6 weeks.
- Home Based: Participants were asked to exercise in their home for 25 minutes 3 times a week for 6 weeks.
Period: Overall Study
Arm/Group | School Based | Home Based
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | School Based | Home Based | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 16 (0.8) | 17 (0.0) | 17 (0.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 9
Primary Disability [Count of Participants; unit: Participants]
  Down Syndrome | 1 | 0 | 1
  Autism Spectrum Disorder (ASD) | 1 | 0 | 1
  Post Cranial Surgery | 1 | 0 | 1
  Attention-Deficit/Hyperactivity Disorder (ADHD) | 1 | 2 | 3
  Cerebral Palsy | 0 | 1 | 1
  Autism Spectrum Disorder (ASD) and Attention-Deficit/Hyperactivity Disorder (ADHD) | 1 | 0 | 1
  Specific Learning Disability (SLD) | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Attendance
Description: The percentage of session attended over the 6 week duration. Values were found by taking the total number of session attended by each group, divided by the total number of session across 6 weeks.
Time Frame: Weeks 1 to 6
Measure: Number; unit: percentage of total sessions attended
Arm/Group | School Based | Home Based
Number analyzed (Participants) | 5 | 4
percentage of total sessions attended | 84.4 | 31.9

2. Primary Outcome: Move Minutes
Description: Average Move minutes obtained per week. Move minutes across the 6 week duration were summed and averaged per group at the given exercise perscription.
Time Frame: Weeks 1 to 6
Measure: Mean (Standard Deviation); unit: Average Move Minutes per week
Arm/Group | School Based | Home Based
Number analyzed (Participants) | 5 | 4
Average Move Minutes per week | 18 (1.41) | 17.25 (18.08)

3. Secondary Outcome: Walking Endurance
Description: Distance (in meters) covered throughout a 6 minute walk.
Time Frame: Week 1 and Week 6
Measure: Mean (Standard Deviation); unit: Meters traveled in 6 minutes
Arm/Group | School Based | Home Based
Number analyzed (Participants) | 5 | 4
Meters traveled in 6 minutes
  Week 1 | 424.61 (107.69) | 473.89 (78.03)
  Week 6 | 442.55 (83.06) | 501.06 (68.32)

4. Secondary Outcome: Hand Grip Strength
Description: Hand grip strength measured via a digital hand dynamometer
Time Frame: Week 1 and Week 6
Measure: Mean (Standard Deviation); unit: Average Kilograms
Arm/Group | School Based | Home Based
Number analyzed (Participants) | 5 | 4
Average Kilograms
  Week 1 Left | 24.2 (10.5) | 25.8 (5.6)
  Week 1 Right | 26.3 (10.8) | 27.3 (5.0)
  Week 6 Left | 23.7 (10.9) | 24.2 (8.3)
  Week 6 Right | 27.1 (13.0) | 28.5 (6.5)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Virtual Reality Exercise Program in Special Physical Education: During normal special physical education hours participants were provided with a virtual reality headset and exercise games. Over 6 weeks they were prescribed to exercise at a moderate intensity 3 times a week for 25 minutes, during their special physical education period.
- Home-based Virtual Reality Exercise Program: Participants were provided with a virtual reality headset and exercise games. Over 6 weeks they were prescribed to exercise at a moderate intensity 3 times a week for 25 minutes at their homes.
Arm/Group | Virtual Reality Exercise Program in Special Physical Education | Home-based Virtual Reality Exercise Program
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT05935982/Prot_SAP_000.pdf